CLINICAL TRIAL: NCT05120700
Title: Effectiveness and Safety of Synovial Tissue and Fat Pad Stromal Vascular Fraction Bioengineering in Patients With Knee Articular Cartilage Injury, Clinical Study Phase I/II
Brief Title: Synovial Tissue and Fat Pad Stromal Vascular Fraction Bioengineering in Patients With Knee Articular Cartilage Injury
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of Sao Paulo General Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 4.285.308
Record Dates: First submitted 2021-10-18; First posted 2021-11-15 (Actual); Last update posted 2021-11-15 (Actual); Status verified 2021-10

CONDITIONS: Cell- and Tissue-Based Therapy; Cartilage Injury; Knee Injuries
Keywords: Tissue engineering; Cell- and Tissue-Based Therapy; Mesenchymal Stem Cells; Cartilage; Knee.
MeSH Terms: conditions — Knee Injuries

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Stromal vascular fraction (Experimental): Treatment of cartilage injury with a tissue engineering construct.The patients will be adults diagnosed with a single, 3 to 6 cm2 full-thickness cartilage lesion, symptomatic and with no improvement with non-operative treatment.
  Interventions: Biological: Synovial Tissue and Fat Pad Stromal Vascular Fraction

INTERVENTIONS:
Biological: Synovial Tissue and Fat Pad Stromal Vascular Fraction — Treatment of cartilage injury with a tissue engineering construct. It will be composed of stromal vascular fraction collected from the synovial membrane and infrapatellar fat of the injured knee, submitted to enzymatic processing in a single surgical time, associated with a collagen scaffold

SUMMARY:
A phase I/II clinical trial (first in human) to assess the effectiveness and safety of the treatment of cartilage injury with a tissue engineering construct composed of stromal vascular fraction collected from the synovial membrane and infrapatellar fat of the injured knee, submitted to enzymatic processing in a single surgical time, associated with a collagen scaffold.

The primary outcomes will be assessed by 3T magnetic resonance imaging, quality of life and knee function questionnaires, in addition to perioperative and post-operative complications. Secondary outcomes will be evaluated by measuring the health resources used to ensure compatibility, reproducibility and generalizability of the technique.

The authors believe that adverse events will be similar to current surgical procedures and that there will be an improvement in knee function scores and quality of life of patients undergoing the procedure.

DETAILED DESCRIPTION:
Introduction: Cartilage injuries affect up to 63% of the population, and can cause pain and important functional limitations. The evolution to osteoarthritis can lead to a worsening of quality of life, in addition to being highly disabling. Osteoarthritis is considered a public healthcare disease with a high economic and social burden without definitive treatment. Despite the various techniques available today, complete regeneration of damaged hyaline cartilage is not possible. For these reasons, cell therapy with mesenchymal cells has received more attention in research due to the relative ease of processing. Synovia and infra-patellar fat-pad are predictable and easily accessible sources during routine arthroscopic procedure, in addition to exhibiting the greatest potential for chondrogenic differentiation between mesenchymal cell donor sites. In a previous pre-clinical translational study (FAPESP - State of São Paulo Government Research Sponsor Agency), The authors' group developed the tissue bioengineering protocol in a large animal model according to the good laboratory practices for in human usage techniques (GMP). After completing this step, The authors now propose the phase I/II clinical trial.

Purpose: The aim of the study is to evaluate effectiveness and safety for the treatment of articular cartilage injuries, with a compound of stromal vascular fraction acquired from the synovia and infrapatellar fat pad of the knee, associated with a collagen scaffold.

Methods: A phase I/II clinical trial (first in human) to assess the safety and efficacy of the treatment of cartilage injury with a tissue engineering construct.

Inclusion criteria: Patients diagnosed with a single, 3 to 6 cm2 full-thickness cartilage lesion, symptomatic and without improvement with non-operative treatment. Age between 18 and 40 years.

Exclusion criteria: any previous surgery to treat the injury, presence of pathology in the contralateral knee or other pathologies that interfere with recovery. Serological tests will be performed for autologous donors, complete serology: HIV, hepatitis C virus, hepatitis B, human T-lymphotropic virus, syphilis and Chagas.

Our institutional ethics committees approved the protocol (local CEP: 4.285.308 and national CAAE: 34798720.5.0000.0068).

The bioengineering construct will be composed of stromal vascular fraction collected from the synovial membrane and infrapatellar fat of the injured knee, submitted to enzymatic processing in a single surgical time, associated with a collagen scaffold (Chondro-Gide, Geistlich, Switzerland). The synovial and adipose tissue are collected through the usual route of the initial surgical incision for cartilage repair, and subsequently centrifuged for 3 minutes.

The isolation of the vascular-stromal fraction will be carried out through enzymatic digestion with collagenase IA. The cell suspension will be centrifuged and the cell button will be suspended in 1 mL of 0.9% saline solution. In one gram of adipose tissue, it is found an average of 2x106 cells, 10% being composed of stromal cells derived from adipocytes.

Demographic data of patients will be collected, as well as data on the frequency of complications in the perioperative, immediate and late postoperative periods. The impact on quality of life and knee function will be assessed by questionnaires. The length of hospital stay, as well as surgical and outpatient care costs, will be documented. The tissue formed after the intervention will be evaluated using the modified 3D MOCART score.

Demographic data will be presented in the form of graphs and tables, as well as the respective frequency distributions of possible complications in the perioperative and postoperative period, and the assessment of economic feasibility. Statistical analyzes will be performed to compare the preoperative and postoperative periods.

To assess the assumption of normal distribution, the Shapiro-Wilk test will be performed, and for the analysis of homogeneity of variances, the Levene test will be performed. In all inferential analyses, a type I error probability (α) of 0.05 will be considered. To evaluate the quantitative variables, Student's t test (or Mann-Whitney test, if the variables do not present normal distribution) or Multivariate Analysis of Variance (MANOVA) will be used. To verify the association between categorical variables, the chi-square association test will be used. For all analyses, the SIGMAPlot 12.5 software (Systat Software, Inc.) will be used.

The authors will also perform the assessment by laboratory characterization of the vascular stromal fraction of mesenchymal stromal cells with two methodologies: flow cytometry immunophenotyping analysis and cell differentiation analysis for osteogenic lineage, previously validated by the research group.

Results:

The primary outcomes will be assessed preoperatively, at 6 and 12 months postoperatively by 3T magnetic resonance imaging (quantity and quality of repair), quality of life and knee function questionnaires, in addition to perioperative and post-operative complications. Secondary outcomes will be evaluated by measuring the health resources used to ensure compatibility, reproducibility and generalizability of the technique.

Hypothesis: The authors believe that adverse events such as pain, bleeding and fever will be similar to current surgical procedures. The authors believe that there will be an improvement in knee function scores and quality of life of patients undergoing the procedure from the non-invasive evaluation by magnetic resonance with good quality cartilage tissue.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with a single, 3 to 6 cm2 full-thickness cartilage lesion, symptomatic and without improvement with non-operative treatment.

Exclusion Criteria:

* Any previous surgery to treat the injury, presence of pathology in the contralateral knee or other pathologies that interfere with recovery. Serological tests will be performed for autologous donors, complete serology: HIV, HCV, HBsAg, anti HBC, HTLV I and II, syphilis and Chagas.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 10 (Estimated)
Dates: Start 2022-04 (Estimated); Primary Completion 2025-04 (Estimated); Study Completion 2025-05 (Estimated)

PRIMARY OUTCOMES:
Cartilage Repair | The primary outcomes will be assessed preoperatively in the allocation date; at 6 months postoperatively; and at 12 months postoperatively
  3T magnetic resonance imaging to evalate quantity and quality of cartilage repair
Visual Analog Score for pain | The primary outcomes will be assessed preoperatively in the allocation date; at 6 months postoperatively; and at 12 months postoperatively
  A patient is asked to indicate his/her perceived pain intensity (most commonly) along a 100 mm horizontal line, and this rating is then measured from the left edge.
International Knee Documentation Committee Questionnaire | The primary outcomes will be assessed preoperatively in the allocation date; at 6 months postoperatively; and at 12 months postoperatively
  The questionnaire looks at 3 categories: symptoms, sports activity, and knee function. The symptoms subscale helps to evaluate things such as pain, stiffness, swelling and giving-way of the knee
Western Ontario and McMaster Universities Osteoarthritis Index | The primary outcomes will be assessed preoperatively in the allocation date; at 6 months postoperatively; and at 12 months postoperatively
  WOMAC evaluates the condition of patients with osteoarthritis of the knee, including pain, stiffness, and physical functioning of the join
Perioperative and post-operative complications | Since hospital admission for the procure until hospital discharge; and monthly after discharge, until 12 months postoperatively
  Assessment of wound infections, pneumonia, cardiovascular and cerebrovascular events, deep vein thrombosis and/or pulmonary embolisms, ICU-admission, hospital readmission and need for complication surgery

SECONDARY OUTCOMES:
Measurement of health resources expenses | Since allocation date; until 12 months postoperatively
  Resources expenses with the procedure to ensure compatibility, reproducibility and generalizability of the technique